CLINICAL TRIAL: NCT03905512
Title: A Study to Compare the Efficacy of SEL-212 to KRYSTEXXA® in Gout Patients Refractory to Conventional Therapy
Brief Title: A Study to Compare the Efficacy of SEL-212 to KRYSTEXXA® in Gout Participants Refractory to Conventional Therapy
Acronym: COMPARE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Selecta Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEL-212/202
Record Dates: First submitted 2019-04-01; First posted 2019-04-05 (Actual); Results first posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Chronic Gout
MeSH Terms: interventions — Pegloticase

STUDY DESIGN:
Masking Description: Assessments of qualitative endpoints will be conducted on an assessor-blinded basis.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SEL-212 (Experimental): Intravenous (IV) infusion of SEL-212 every 28 days for up to 6 infusions
  Interventions: Drug: SEL-212
- KRYSTEXXA (Active Comparator): IV infusion of KRYSTEXXA® according to the manufacturer's prescribing information every 14 days for up to 12 infusions
  Interventions: Drug: KRYSTEXXA®

INTERVENTIONS:
Drug: SEL-212 — Administered as specified in the treatment arm
  Arms: SEL-212
Drug: KRYSTEXXA® — Administered as specified in the treatment arm
  Other Names: Pegloticase
  Arms: KRYSTEXXA

SUMMARY:
This is a randomized, parallel-arm, multicenter study to compare the safety and efficacy profiles of SEL-212 and KRYSTEXXA®. Participants will be randomized 1:1 to receive treatment with SEL-212 or KRYSTEXXA® for 6 months. Efficacy assessments, as measured by serum uric acid (SUA) levels, will be conducted at intervals that are appropriate to determine treatment effect differences. Safety will be monitored throughout the study.

DETAILED DESCRIPTION:
This is a randomized, parallel-arm, multicenter study to compare the safety and efficacy profiles of SEL-212 and KRYSTEXXA®. Participants will be randomized 1:1 to receive treatment with SEL-212 [a combination of pegadricase (SEL-037) and ImmTOR (SEL-110)] or KRYSTEXXA® for 6 months.

Study participants in the SEL-212 arm will receive study drug every 28 days for a total of up to 6 infusions of SEL-212. Study participants in the KRYSTEXXA® arm will receive study drug according to the manufacturer's prescribing information, i.e., every 14 days for a total of up to 12 infusions of KRYSTEXXA®.

Efficacy assessments, as measured by SUA levels, will be conducted at intervals that are appropriate to determine treatment effect differences. Safety will be monitored throughout the study.

ELIGIBILITY:
Key Inclusion Criteria:

1. History of symptomatic gout defined as:

   1. ≥ 3 gout flares within 18 months of Screening or
   2. Presence of ≥ 1 tophus or
   3. Current diagnosis of gouty arthritis
2. At the Screening Visit: male age 21 - 80 years, inclusive, or female of non-childbearing potential age 21-80 years, inclusive, where non-childbearing potential is defined as:

   1. > 6 weeks after hysterectomy with or without surgical bilateral salpingooperhectony or
   2. Post-menopausal (> 24 months of natural amenorrhea)
3. Has at the Screening Visit SUA ≥ 7 mg/dL, with chronic refractory gout defined as having failed to normalize SUA and whose signs and symptoms are inadequately controlled with xanthine oxidase inhibitors at the medically appropriate dose or for whom these drugs are contraindicated;
4. Willing to provide written informed consent prior to the conduct of any study specific procedures;
5. Understands and is willing and able to comply with study requirements, including the schedule of follow-up visits

Key Exclusion Criteria:

1. Prior exposure to any experimental or marketed uricase (e.g., pegloticase [Krystexxa®], pegadricase [SEL-037], rasburicase [Elitek, Fasturtec]);
2. History of anaphylaxis or severe allergic reactions to medications;
3. History of any allergy to pegylated products
4. Drugs known to interact with Rapamune cannot be used during the trial;
5. Uncontrolled diabetes;
6. Glucose-6-phosphate dehydrogenase (G6PD) deficiency;
7. Uncontrolled hypertension;
8. Participants whose arrhythmia is unstable on current treatment;
9. History of coronary artery disease, including myocardial infarction or unstable angina, within the last 6 months;
10. Congestive heart failure;
11. History of hematological disorders within 1 year or autoimmune disorders, is immunosuppressed or immunocompromised;
12. Has received an inactivated vaccine in the previous 3 months or has received a live virus vaccine in the previous 6 months;
13. Is planning to receive any vaccination or live virus vaccination during the study;

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 170 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Selecta Biosciences, Inc.
Locations (42):
- United States (42):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Arizona Arthritis & Rheumatology Research, PLLC, Sun City, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Medvin Clinical Research, Covina, California
  - Valerius Medical Group and Research Center of Greater Long Beach, Inc., Los Alamitos, California
  - Arthritis Care and Research Center, Poway, California
  - MD Strategies Research Centers, San Diego, California
  - Clinical Research of West Florida, Clearwater, Florida
  - QPS-Medical Research Assoc LLC, Miami, Florida
  - Well Pharma Medical Research Corp., Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Accelerated Enrollment Solutions (AES), Orlando, Florida
  - Rheumatology Associates of Central Florida, PA, Orlando, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Advent Health Group Multispecialty at Habana and Bruce B. Downs, Tampa, Florida
  - Arthritis Center of North Georgia, Gainesville, Georgia
  - Better Health Clinical Research, Inc., Newnan, Georgia
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Great Lakes Clinical Trials, Chicago, Illinois
  - L-MARC Research Center, Louisville, Kentucky
  - Klein & Associates, M.D., P.A., Cumberland, Maryland
  - Klein & Associates, M.D., P.A., Hagerstown, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - University Hospital, Ann Arbor, Michigan
  - Elite Clinical Research, LLC, Jackson, Mississippi
  - TEST, Blue Springs, Missouri
  - NYU Langone Ambulatory Care Brooklyn Heights, Brooklyn, New York
  - DJL Clinical Research, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cape Fear Arthritis Care PLLC, Leland, North Carolina
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Arthritis & Rheumatology Center of Oklamhoma, PLLC, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading, LLC, Wyomissing, Pennsylvania
  - West Tennessee Research Institute, LLC, Jackson, Tennessee
  - Amarillo Center for Clinical Research, Amarillo, Texas
  - Austin Regional Clinic, Austin, Texas
  - Tekton Research, Austin, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Southwest Rheumatology Research, LLC, Mesquite, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baraf HSB, Khanna PP, Kivitz AJ, Strand V, Choi HK, Terkeltaub R, Dalbeth N, DeHaan W, Azeem R, Traber PG, Keenan RT. The COMPARE head-to-head, randomized controlled trial of SEL-212 (pegadricase plus rapamycin-containing nanoparticle, ImmTOR) versus pegloticase for refractory gout. Rheumatology (Oxford). 2024 Apr 2;63(4):1058-1067. doi: 10.1093/rheumatology/kead333. PMID 37449908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled across clinical sites in the United States.
Groups:
- SEL-212: Participants received SEL-212 via intravenous (IV) infusion every 28 days for up to 6 months
- KRYSTEXXA: Participants received KRYSTEXXA® according to the manufacturer's prescribing information every 14 days for up to 6 months
Period: Overall Study
Arm/Group | SEL-212 | KRYSTEXXA
Started | 83 | 87
Received At Least 1 Dose of Study Drug | 83 | 87
Completed | 62 | 70
Not Completed | 21 | 17
Not completed — Withdrawal by Subject | 9 | 8
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 4 | 3
Not completed — Other than Specified | 7 | 4

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) set included all randomized participants.
Groups:
- SEL-212: Participants received SEL-212 via IV infusion every 28 days for up to 6 months
- Total: Total of all reporting groups
Arm/Group | SEL-212 | KRYSTEXXA | Total
Number analyzed (Participants) | 83 | 87 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (11.47) | 52.0 (10.43) | 52.3 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 78 | 85 | 163
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 21 | 36
  Not Hispanic or Latino | 68 | 66 | 134
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 16 | 16 | 32
  White | 62 | 69 | 131
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serum Uric Acid (SUA) Reduction of < 6 mg/dL for at Least 80% of the Time
Description: The average of the data collected during Month 3 and Month 6 was reported.
Time Frame: Up to Month 6
Population: ITT set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | SEL-212 | KRYSTEXXA
Number analyzed (Participants) | 83 | 87
Participants | 44 | 40
Statistical Analysis 1: Comparison: SEL-212 vs KRYSTEXXA; Test type: Superiority — Statistical significance was tested at a level of 0.05; p = 0.181, Cochran-Mantel-Haenszel

2. Secondary Outcome: Number of Participants With SUA Reduction of < 6 mg/dL for At Least 80% of the Time During Month 6
Time Frame: Month 6
Population: ITT set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | SEL-212 | KRYSTEXXA
Number analyzed (Participants) | 83 | 87
Participants | 45 | 41

3. Secondary Outcome: Number of Participants With SUA Reduction of < 6 mg/dL for 100% of the Time During Month 6
Time Frame: Month 6
Population: ITT set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | SEL-212 | KRYSTEXXA
Number analyzed (Participants) | 83 | 87
Participants | 38 | 36

4. Secondary Outcome: Quality of Life (QoL) as Assessed by Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Scale
Description: Eight categories were assessed by the HAQ-DI: 1) dressing and grooming, 2) arising, 3) eating, 4) walking, 5) hygiene, 6) reaching, 7) gripping, and 8) common daily activities. There were 2 or 3 questions for each category.
  Scoring within each category was on a 4-point Likert scale from 0 (without any difficulty) to 3 (unable to do). The score given to each section was the worst (highest) score within the section. The HAQ-DI total score was calculated if 6 or more sections were available. The average of the 8 category scores was reported as the HAQ-DI total score on a scale of 0 to 3. Reduction from baseline, and lower scores indicated better QoL.
Time Frame: Baseline to End of Month 3, Baseline to End of Month 6
Population: ITT set included all randomized participants. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure and 'Number analyzed' = participants evaluable at the specified timeframe.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SEL-212 | KRYSTEXXA
Number analyzed (Participants) | 82 | 83
score on a scale
  Baseline | 0.78 (0.774) | 0.79 (0.834)
  Change at End of Month 3: number analyzed (Participants) | 61 | 66
  Change at End of Month 3 | -0.14 (0.725) | -0.10 (0.795)
  Change at End of Month 6: number analyzed (Participants) | 59 | 65
  Change at End of Month 6 | 0.04 (0.723) | -0.12 (0.739)

5. Secondary Outcome: QoL as Assessed by Change From Baseline in Provider Global Assessment of Disease Activity (PrGA) Scale
Description: The PrGA was administered to assess the severity of the participant's disease on a scale from 0 (participant feels "very well") to 100 (participant feels "very poor"). Reduction from baseline, and lower scores indicated less severe disease.
Time Frame: Baseline to End of Month 3, Baseline to End of Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SEL-212 | KRYSTEXXA
Number analyzed (Participants) | 78 | 81
score on a scale
  Baseline | 42.8 (26.65) | 40.5 (28.62)
  Change at End of Month 3: number analyzed (Participants) | 60 | 67
  Change at End of Month 3 | -20.9 (25.38) | -15.8 (32.97)
  Change at End of Month 6: number analyzed (Participants) | 51 | 62
  Change at End of Month 6 | -24.6 (24.87) | -22.0 (29.37)

6. Secondary Outcome: QoL as Assessed by Change From Baseline in Short Form Health Survey 36 (SF-36) Scale
Description: The SF-36 is a 36-item questionnaire to assesses a participant's health status using 8 health concepts: limitations in physical activities because of health problems; limitations in social activities because of physical or emotional problems; limitations in usual role activities because of physical health problems; bodily pain; general mental health (psychological distress and well-being); limitations in usual role activities because of emotional problems; vitality (energy and fatigue); and general health perceptions.
  The mental component reports the average of all the emotionally relevant items and the physical component reports the average of all the physical relevant items. Each component is directly transformed into a 0 to 100 scale on the assumption that each question carries equal weight. A score of 0 is equal to maximum disability, and a score of 100 indicates no disability. Median change can range from -100 to 100. A positive median change indicated an improved outcome.
Time Frame: Baseline to End of Month 3, Baseline to End of Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SEL-212 | KRYSTEXXA
Number analyzed (Participants) | 81 | 84
score on a scale
  Physical Component Scores at Baseline | 43.822 (10.9976) | 43.345 (11.2714)
  Change in Physical Component Scores at End of Month 3: number analyzed (Participants) | 60 | 69
  Change in Physical Component Scores at End of Month 3 | 3.323 (9.9242) | 5.768 (9.0712)
  Change in Physical Component Scores at End of Month 6: number analyzed (Participants) | 59 | 66
  Change in Physical Component Scores at End of Month 6 | 5.881 (9.0453) | 7.448 (8.3909)
  Mental Component Scores at Baseline | 51.977 (8.4731) | 53.386 (9.3171)
  Change in Mental Component Scores at End of Month 3: number analyzed (Participants) | 60 | 69
  Change in Mental Component Scores at End of Month 3 | 0.381 (6.7469) | 1.229 (7.6445)
  Change in Mental Component Scores at End of Month 6: number analyzed (Participants) | 59 | 66
  Change in Mental Component Scores at End of Month 6 | 1.516 (6.4824) | -0.322 (8.0626)

7. Secondary Outcome: Number of Participants With Gout Flares Per 3-Month Period
Time Frame: Month 1 to Month 3, Month 4 to Month 6
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | SEL-212 | KRYSTEXXA
Number analyzed (Participants) | 83 | 87
Participants
  Month 1 to Month 3 | 50 | 42
  Month 4 to Month 6: number analyzed (Participants) | 68 | 75
  Month 4 to Month 6 | 16 | 15

8. Secondary Outcome: Number of Gout Flares Per 3-Month Period
Time Frame: Month 1 to Month 3, Month 4 to Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: number of flares
Arm/Group | SEL-212 | KRYSTEXXA
Number analyzed (Participants) | 83 | 87
number of flares
  Month 1 to Month 3 | 1.1 (1.16) | 0.8 (1.24)
  Mont 4 to Month 6: number analyzed (Participants) | 68 | 75
  Mont 4 to Month 6 | 0.2 (0.56) | 0.3 (1.15)

9. Secondary Outcome: Change From Baseline in Number of Tender Joints
Time Frame: Baseline to End of Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: number of tender joints
Arm/Group | SEL-212 | KRYSTEXXA
Number analyzed (Participants) | 82 | 87
number of tender joints
  Baseline | 5.2 (8.81) | 4.1 (7.49)
  Change at End of Month 6: number analyzed (Participants) | 56 | 67
  Change at End of Month 6 | -2.4 (8.98) | -2.7 (6.93)

10. Secondary Outcome: Change From Baseline in Number of Swollen Joints
Time Frame: Baseline to End of Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: number of swollen joints
Groups:
- KRYSTEXXA: Participants received KRYSTEXXA® according to the manufacturer's prescribing information every 14 days up to 6 months
Arm/Group | SEL-212 | KRYSTEXXA
Number analyzed (Participants) | 82 | 87
number of swollen joints
  Baseline | 3.0 (5.39) | 3.7 (6.64)
  Change at End of Month 6: number analyzed (Participants) | 56 | 67
  Change at End of Month 6 | -1.6 (5.51) | -1.9 (8.38)

ADVERSE EVENTS:
Time Frame: Up to 7 months
Description: Safety Set included all participants who received the study drug.
Arm/Group | SEL-212 | KRYSTEXXA
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/87
Serious Adverse Events (participants affected / at risk) | 7/83 | 8/87
Other Adverse Events (participants affected / at risk) | 60/83 | 53/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SEL-212 (N=83) | KRYSTEXXA (N=87)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Coronavirus infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Hypertensive emergency (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SEL-212 (N=83) | KRYSTEXXA (N=87)
Diarrhoea (Gastrointestinal disorders) | 5 | 0
Infusion Related reaction (Injury, poisoning and procedural complications) | 13 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 6
Headache (Nervous system disorders) | 6 | 0
Hematuria (Renal and urinary disorders) | 5 | 0
Hypertension (Vascular disorders) | 6 | 5
Gout (Metabolism and nutrition disorders) | 50 | 44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT03905512/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT03905512/SAP_001.pdf